CLINICAL TRIAL: NCT01044745
Title: Rituximab For Prevention Of Acute Graft-Versus-Host Disease (GVHD) After Unrelated Donor Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Rituximab in Preventing Acute Graft-Versus-Host Disease in a Donor Stem Cell Transplant for Hematologic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed to accrual for safety related to the frequency of BK infections.
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0083-09-FB; NCI-2009-01552 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Blastic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Graft Versus Host Disease; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage I Small Lymphocytic Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Lymphoma, Extranodal NK-T-Cell; Blast Crisis; Graft vs Host Disease; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; Mycophenolic Acid; Tacrolimus; Antilymphocyte Serum; thymoglobulin; Therapeutics; Cyclophosphamide; fludarabine phosphate; Busulfan; Whole-Body Irradiation; Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Rituximab and allogeneic HCT transplant) (Experimental): CONDITIONING REGIMEN: Patients receive one of the following conditioning regimens as per the transplant physician: cyclophosphamide and TBI; targeted busulfan and fludarabine; reduced-dose busulfan and fludarabine; or fludarabine and TBI.
  GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive rituximab IV on days -6, 1, 8, and 15 and anti-thymocyte globulin IV over 6-8 hours on days -3 to -1. Patients also receive tacrolimus IV continuously and then PO beginning on day -1 and continuing until day 150 followed by a taper until day 180 and mycophenolate mofetil PO or IV twice daily on days -1 to 60.
  TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0.
  Interventions: Drug: rituximab; Drug: mycophenolate mofetil; Drug: tacrolimus; Drug: anti-thymocyte globulin; Procedure: allogeneic hematopoietic stem cell transplantation; Other: laboratory biomarker analysis; Biological: graft versus host disease prophylaxis/therapy; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: busulfan; Radiation: total-body irradiation; Biological: graft-versus-tumor induction therapy; Biological: immunosuppressive therapy

INTERVENTIONS:
Drug: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: mycophenolate mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Drug: tacrolimus — Given IV
  Other Names: FK 506; Prograf
Drug: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Procedure: allogeneic hematopoietic stem cell transplantation — Stem cell transplant
Other: laboratory biomarker analysis — Correlative studies
Biological: graft versus host disease prophylaxis/therapy — Undergo graft versus host disease prophylaxis/therapy
  Other Names: prophylaxis/therapy, graft versus host disease; prophylaxis/therapy, GVHD
Drug: cyclophosphamide — Given PO or IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Biological: graft-versus-tumor induction therapy — Undergo graft-versus-tumor induction therapy
  Other Names: graft versus host disease induction; graft versus tumor induction
Biological: immunosuppressive therapy — Undergo immunosuppressive therapy
  Other Names: immunosuppression

SUMMARY:
This phase II trial is studying how well rituximab works in preventing acute graft-versus-host disease (GVHD) in patients undergoing a donor stem cell transplant for hematologic cancer. Giving chemotherapy and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving a monoclonal antibody, rituximab, together with anti-thymocyte globulin, tacrolimus, and mycophenolate mofetil before and after the transplant may stop this from happening

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the incidence of grade II-IV acute GVHD at day 100 after matched unrelated donor allogeneic hematopoietic cell transplantation (HCT) when incorporating rituximab in the conditioning regimen.

SECONDARY OBJECTIVES:

I. To determine the day 100 transplant related mortality after matched unrelated donor allogeneic HCT when incorporating rituximab in the conditioning regimen.

II. To determine overall survival (OS) and disease-free survival (DFS) after matched unrelated donor allogeneic HCT when incorporating rituximab in the conditioning regimen.

III. To determine the cumulative incidence of infectious complications at day 100 after matched unrelated donor HCT when incorporating rituximab in the conditioning regimen.

IV. To determine the effect of rituximab addition to the conditioning regimen on recovery of T regulatory (T-reg) cells, and to determine the effect of T-cell, including T-reg, number in the stem cell product and at day 30 on the incidence of grade II-IV acute GVHD (aGVHD) and the cumulative infectious complications at day 100.

V. To determine the effect of rituximab addition to the conditioning regimen on antigen presenting myeloid cell recovery, and to determine the effect of dendritic cell subset DC1, DC2 and myeloid-derived suppressor cells (MDSC), number in the stem cell graft and at day +30 on the incidence of acute GVHD grade II-IV and the cumulative incidence of infectious complications at day 100.

OUTLINE:

CONDITIONING REGIMEN: Patients receive one of the following conditioning regimens as per the transplant physician: cyclophosphamide and total-body irradiation (TBI); targeted busulfan and fludarabine; reduced-dose busulfan and fludarabine; or fludarabine and TBI.

GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive rituximab intravenously (IV) on days -6, 1, 8, and 15 and anti-thymocyte globulin IV over 6-8 hours on days -3 to -1. Patients also receive tacrolimus IV continuously and then orally (PO) beginning on day -1 and continuing until day 150 followed by a taper until day 180 and mycophenolate mofetil PO or IV twice daily on days -1 to 60.

TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0.

Patients are followed up periodically for 100 days after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myelogenous leukemia (CML) in accelerated phase or blast crisis, chronic lymphocytic leukemia (CLL), Non-Hodgkin lymphoma (NHL), myelodysplastic syndromes (MDS) (intermediate-2 or high-risk disease by International Pelvic Pain Society [IPPS])
* Patients with AML, ALL, or MDS scheduled for myeloablative conditioning should have =< 10% blasts in bone marrow or peripheral blood at the start of conditioning
* Patients with AML, ALL, or CML scheduled for reduced intensity conditioning or non-myeloablative conditioning should be in complete morphologic remission at the start of conditioning (residual disease by flow cytometry or cytogenetics and/or incomplete recovery of neutrophil or platelet count are acceptable)
* Patients with CLL or NHL scheduled for reduced intensity or non-myeloablative conditioning should have no evidence of bulky disease (> 50% bone marrow involvement or masses > 10 cm) at the start of conditioning
* Fulfills all pulmonary, cardiac, renal, and hepatic criteria for standard-of-care matched unrelated donor (MUD) allogeneic HCT
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after stem cell transplantation
* Adequately matched unrelated donor available
* Written informed consent; written informed consent of the unrelated donor is required to participate in the optional studies

Exclusion Criteria:

* Patient or donor infected with human immunodeficiency virus (HIV)
* Patient or donor with history of hepatitis B or C and/or positive serology consistent with previous hepatitis B or C infection (patients and/or donor who received Hepatitis B vaccination are acceptable)
* Patient or donor with active hepatitis B or C and/or detectable viral ribonucleic acid (RNA)
* More than 20,000 circulating CD20+ cells/uL
* Treatment with rituximab for any reason in the 12 months preceding HCT
* Patient scheduled for cord blood transplantation
* Presence of active uncontrolled infection at start of conditioning
* Presence of active central nervous system (CNS) disease (history of adequately treated CNS disease is acceptable)
* Presence of uncontrolled psychiatric disorder
* Patient unable to give informed consent
* Unrelated donor products received from the Deutsche Knochenmarkspenderdatei (DKMS) Registry are not eligible for the optional study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12-10 (Actual); Primary Completion 2012-12-19 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bociek, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Rituximab and Allogeneic HCT Transplant): CONDITIONING REGIMEN: Cyclophosphamide and TBI; targeted busulfan and fludarabine; reduced-dose busulfan and fludarabine; or fludarabine and TBI.
  GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Rituximab IV days -6, 1, 8, and 15 and anti-thymocyte globulin IV over 6-8 hours on days -3 to -1. Tacrolimus IV continuously and then PO beginning on day -1 and continuing until day 150 followed by a taper until day 180 and mycophenolate mofetil PO or IV twice daily on days -1 to 60.
  TRANSPLANTATION: Allogeneic hematopoietic stem cell transplantation on day 0.
  laboratory biomarker analysis: Correlative studies
  graft versus host disease prophylaxis/therapy: Undergo graft versus host disease prophylaxis/therapy
  cyclophosphamide: Given PO or IV
  fludarabine phosphate: Given IV
  busulfan: Given IV
  total-body irradiation: Undergo TBI
  graft-versus-tumor induction therapy: Undergo graft-versus-tumor induction therapy
  immunosuppressive therapy: Undergo immunosuppressive therapy
Period: Overall Study
Arm/Group | Treatment (Rituximab and Allogeneic HCT Transplant)
Started | 20
Completed | 18
Not Completed | 2
Not completed — Ineiligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Rituximab and Allogeneic HCT Transplant)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 39 [21 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grades II-IV Acute GVHD
Description: Determined with death as a competing risk. Defined and staged using the 1994 consensus conference modifications of the Glucksberg criteria.
Time Frame: At day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab and Allogeneic HCT Transplant)
Number analyzed (Participants) | 20
Participants | 16

2. Secondary Outcome: Event-free Survival
Description: Estimated using Kaplan-Meier estimator.
Time Frame: From the date of transplant with relapse/progression or death as censored events, up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Rituximab and Allogeneic HCT Transplant)
Number analyzed (Participants) | 18
months | 12 [6 to 18]

3. Secondary Outcome: Overall Survival
Description: Estimated using Kaplan-Meier estimator.
Time Frame: From the date of transplant with death from any cause as a censored event, up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Rituximab and Allogeneic HCT Transplant)
Number analyzed (Participants) | 18
months | 12 [9 to 18]

4. Secondary Outcome: Transplant-related Mortality (TRM)
Description: Transplant-related mortality (TRM) defined as any mortality after transplantation except mortality from relapsed disease - Reported as a simple percentage.
Time Frame: At day 100
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Rituximab and Allogeneic HCT Transplant): CONDITIONING REGIMEN: Patients receive one of the following conditioning regimens as per the transplant physician: cyclophosphamide and TBI; targeted busulfan and fludarabine; reduced-dose busulfan and fludarabine; or fludarabine and TBI.
  GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive rituximab IV on days -6, 1, 8, and 15 and anti-thymocyte globulin IV over 6-8 hours on days -3 to -1. Patients also receive tacrolimus IV continuously and then PO beginning on day -1 and continuing until day 150 followed by a taper until day 180 and mycophenolate mofetil PO or IV twice daily on days -1 to 60.
  TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0.
  rituximab: Given IV
  mycophenolate mofetil: Given IV or PO
  tacrolimus: Given IV
  anti-thymocyte globulin: Given IV
  allogeneic hematopoietic stem cell transplantation
  laboratory biomarker analysis: Correlative studies
  graft versus host disease prophyla
Arm/Group | Treatment (Rituximab and Allogeneic HCT Transplant)
Number analyzed (Participants) | 18
Participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Rituximab and Allogeneic HCT Transplant)
All-Cause Mortality (participants affected / at risk) | 5/20
Serious Adverse Events (participants affected / at risk) | 10/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Rituximab and Allogeneic HCT Transplant) (N=20)
Diarrhea (Gastrointestinal disorders) | 3 (3) — Diarrhea
vomiting (Gastrointestinal disorders) | 1 (1) — vomiting
anorexia (Gastrointestinal disorders) | 1 (1)
pneumonitis (Infections and infestations) | 3 (3)
sepsis (Infections and infestations) | 3 (3)
acute kidney injury (Renal and urinary disorders) | 3 (3)
mucositis oral (Gastrointestinal disorders) | 1 (1)
Immune system disorders-other (Immune system disorders) | 2 (2) — graft-versus-host disease
ileus (Gastrointestinal disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
cystitis (Infections and infestations) | 3 (3) — BK virus cystitis
hematuria (Renal and urinary disorders) | 1 (1)
thrombotic event (Hepatobiliary disorders) | 1 (1) — hepatic veno-occlusive disease
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Rituximab and Allogeneic HCT Transplant) (N=20)
Hypokalemia (Metabolism and nutrition disorders) | 7 (15)
Hyponatremia (Metabolism and nutrition disorders) | 5 (6)
Rash (Infections and infestations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (14)
creatinine increased (Investigations) | 1 (1)
Infection and infestation - Other (Infections and infestations) | 1 (1) — Parvovirus
Sepsis (Infections and infestations) | 5 (8)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) — an ANC <1000/mm3 and a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour.
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) — A disorder characterized by redness, marked discomfort, swelling, and tingling in the palms of the hands or the soles of the feet.
Ascites (Gastrointestinal disorders) | 1 (1) — disorder characterized by accumulation of serous or hemorrhagic fluid in the peritoneal cavity.
Skin infection (Infections and infestations) | 1 (1) — cellulitis
sinusitis (Infections and infestations) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
Lung infection (Infections and infestations) | 2 (2) — pneumonia
Weight loss (Investigations) | 1 (1) — Failure to thrive
dehydration (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Mucositis - oral (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (13)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Immune-system disorders- Other (Immune system disorders) | 2 (3) — GVHD -gut
blood bilirubin increased (Investigations) | 2 (2)
Alanin amintransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase (Investigations) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) — deep vein thrombosis
Altered mental status (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No